CLINICAL TRIAL: NCT04733443
Title: A Prospective, Multicenter, Non-inferior, Randomized Controlled Clinical Trial Comparing the Safety and Efficacy of Sequent ® Please Neo With Biolimus-released Coronary Balloon Catheter in the Treatment of Coronary Stent Restenosis
Brief Title: The Safety and Efficacy of Biolimus in the Treatment of Patients With in Stent Restenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: JW Medical Systems Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JW-BA9-ISR-202001
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biolimus (Experimental): BA9 Drug-eluting Coronary Artery Balloon Catheter Length: 10 / 15 / 20 / 25 / 30 / 35 / 40 /45mm Diameter: 2.0/2.25/2.5/2.75/3.0/3.5/4.0 mm
  Interventions: Device: Biolimus
- SeQuent® Please Neo (Active Comparator): paclitaxel released coronary balloon catheters Length: 10 / 15 / 20 / 25 / 30 / 35 / 40 mm Diameter: 2.0/2.25/2.5/2.75/3.0/3.5/4.0 mm
  Interventions: Device: SeQuent® Please Neo

INTERVENTIONS:
Device: Biolimus — 140 patients who met the inclusion/exclusion criteria for in-stent restenosis were enrolled and assigned to the Biolimus treatment group
  Arms: Biolimus
Device: SeQuent® Please Neo — 140 patients who met the inclusion/exclusion criteria for in-stent restenosis were enrolled and assigned to the SeQuent® Please Neo treatment group
  Arms: SeQuent® Please Neo

SUMMARY:
This study consisted of a randomized controlled trial group and a long balloon observation group.

In the randomized control group, 280 subjects with in-stent restenosis were planned to be recruited and randomly assigned to the test group and the control group in a 1:1 ratio; 30 consecutive subjects will be enrolled in the long balloon observation group, using graceful molimus release coronary balloon catheter with length of 45mm; All 310 subjects were followed up at baseline, surgery, discharge, 1 month after surgery, 6 months after surgery, 9 months after surgery, 1, 2 and 3 years after surgery, and angiography was performed at 9 months after surgery.

DETAILED DESCRIPTION:
This study consisted of a randomized controlled trial group and a long balloon observation group.

In the randomized control group, 280 subjects with in-stent restenosis were planned to be recruited and randomly assigned to the test group and the control group in a 1:1 ratio; 30 consecutive subjects will be enrolled in the long balloon observation group, using graceful molimus release coronary balloon catheter with length of 45mm; All 310 subjects were followed up at baseline, surgery, discharge, 1 month after surgery, 6 months after surgery, 9 months after surgery, 1, 2 and 3 years after surgery, and angiography was performed at 9 months after surgery.

The primary endpoint was late lumen loss at 9 months.

The study will enroll 310 subjects. The sample size determination process is as follows:

Randomized controlled trial group:

A prospective, multicenter, randomized, controlled, non-inferior clinical trial design was used with the primary endpoint of intrasegonal LLL at 9 months postoperatively. Sample size was calculated according to the following assumptions:

1) According to previous clinical studies, the LLL of the segment 9 months after paclitaxel release coronary catheter (Sequent Please) was 0.46±0.48mm[1] and 0.46±0.51mm[2]. 2) In this study, it was estimated that the mean LLL in the lesion segment of the experimental group and the control group 9 months after surgery was 0.46mm, and the standard deviation was 0.50mm. 3) The clinically acceptable non-infertility threshold was 0.195mm. When the significance level of the statistical test was set as one-sided 2.5% and the assurance level was set as 80%, they were randomly divided into groups at a ratio of 1:1. 4) Considering the abscission rate of 25% (at the same time considering the early withdrawal from the group caused by other reasons and the random setting), 280 patients were finally enrolled, including 140 in the experimental group and 140 in the control group.

Long balloon observation group:

Because the maximum length of Sequent ® Please Neo in the control group was 40mm, subjects suitable for 45mm long balloon could not be randomly enrolled in the randomized controlled trial group. Therefore, this observation group was selected with a sample size of 30 cases.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years ≤ subject age ≤80 years;
* 2. Stable angina pectoris, acute coronary syndrome, old myocardial infarction or proven asymptomatic myocardial ischemia;
* 3. Subjects have no contraindications to coronary revascularization (PCI or CABG); -4. Subjects agreed to receive clinical follow-up at discharge, 1 month, 6 months, 9 months, 1 year, 2 years and 3 years after surgery, and angiographic follow-up at 9 months after surgery;
* 5. Subjects can understand the purpose of the study and have sufficient compliance with the study protocol. And willing to sign the informed consent and accept the risks and benefits stated in the informed consent.

Exclusion Criteria:

* 1. Patients with any myocardial infarction within 1 week, or patients whose myocardial enzyme CK or CK-MB has not returned to normal although myocardial infarction has occurred for more than 1 week;
* 2. Patients with severe congestive heart failure (NYHA IV) or severe valvular heart disease;
* 3. Female patients who are planning or are pregnant (or breastfeeding);
* 4. Patients with severe renal failure with creatinine >2.0 mg/dL (177 mol/L);
* 5. Left ventricular ejection fraction <30%;
* 6. Coagulation disorders, platelet count <100×109/ L;
* 7. Patients with cardiogenic shock;
* 8. Patients with concomitant diseases requiring cytoinhibitor or radiotherapy;
* 9. Patients who are known to be allergic to aspirin, clopidogrel, Gracilis, ticagrelor, heparin, contrast agent, paclitaxel, or have contraindications to aspirin, clopidogrel, or Ticagrelor;
* 10. Patients with bleeding constitution or a history of cerebral hemorrhage, active digestive ulcer, or gastrointestinal bleeding in the past 6 months will be restricted or prohibited to use anticoagulant therapy or anticoagulant drugs;
* 11. Patients with a life expectancy of less than 1 year or with underlying factors of difficult clinical follow-up;
* 12. Patients who are participating in any other clinical trial;
* 13. For other reasons, the researchers considered the patients unsuitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2025-02-18 (Estimated)

PRIMARY OUTCOMES:
The late lumen loss | 9 months
  Segmental late lumen loss of target lesions 9 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, Ph.D, Principal Investigator — The First Medical Center of the PLA General Hospital
Locations (1):
- The First Medical Center of the PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Gao L, Qin Q, Zhang J, Jia S, Wu M, He Y, Fu G, Liu J, Chen H, Tong Q, Yu Z, An J, Qiu C, Xu B, Cao Y, Wang C, Ma G. Biolimus-coated versus paclitaxel-coated balloons for coronary in-stent restenosis (BIO ASCEND ISR): a randomised, non-inferiority trial. EuroIntervention. 2024 Jul 1;20(13):e806-e817. doi: 10.4244/EIJ-D-24-00295. PMID 38742581